CLINICAL TRIAL: NCT05426408
Title: Stockholm Myocardial Infarction with Nonobstructive Coronaries Study 3 - Pilot Study of Prevalence of Coronary Microvascular Dysfunction in Myocardial Infarction with Nonobstructive Coronary Arteries
Brief Title: Stockholm Myocardial Infarction with Nonobstructive Coronaries Study 3
Acronym: SMINC-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Per Tornvall, Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SMINC-3
Record Dates: First submitted 2022-06-10; First posted 2022-06-22 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-10

CONDITIONS: Myocardial Infarction with Nonobstructive Coronary Arteries
MeSH Terms: conditions — MINOCA

STUDY DESIGN:
Intervention Model Description: Patients will be their own controls
Masking Description: The investigators who will perform the evaluation of the CMR investigations will be blinded to all clinical data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with MINOCA undergoing CMR (Other): Patients will be their own controls
  Interventions: Diagnostic Test: Cardiac magnetic resonance imaging to study coronary microvascular dysfunction

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance imaging to study coronary microvascular dysfunction — Myocardial perfusion mapping will be investigated after administration of adenosine

SUMMARY:
The present pilot study will investigate the prevalence of CMD in an unselected cohort of patients with the working diagnosis MINOCA and to study if the diagnostic yield can be improved by adding adenosine to the CMR investigation. Patient will be their own controls.

ELIGIBILITY:
Inclusion Criteria:

* a suspected diagnosis of MINOCA or takotsubo syndrome with coronary angiography without diameter stenosis ≥50%
* age 35-80 years
* reading and writing proficiency in Swedish

Exclusion Criteria:

* Claustrofobia
* Arrythmia and/or pacemaker (atrial fibrillation and AV-block I- III)
* Asthma or severe chronic obstructive lung disease
* eGFR < 30 ml/min
* spontaneous coronary artery dissection
* acute pulmonary embolism
* acute myocardial infarction type 2
* cardiomyopathy other than takotsubo syndrome
* a previous myocardial infarction due to CAD

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | Through investigation completion, usually 2 hours
  To increase the diagnostic yield of CMR imaging in MINOCA as a working diagnosis

SECONDARY OUTCOMES:
Prevalence of CMD in MINOCA | Through investigation completion, usually 2 hours
  To determine the proportion of patients with the working diagnosis of MINOCA who have CMD.
Prevalence of CMD in different final MINOCA diagnoses | Through investigation completion, usually 2 hours
  To study the proportions of CMD in patients with a CMR imaging diagnosis of myocardial infarction, Takotsubo, respectively myocarditis and compare them with the results from a healthy control group
Angina pectoris | 3 Months
  To investigate the occurrence of angina pectoris before inclusion and after 3 months and relate it to CMD

CONTACTS AND LOCATIONS:
Overall Officials: Per Tornvall, MD, Principal Investigator — Karolinska Instítutet
Locations (1):
- Per Tornvall, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No